CLINICAL TRIAL: NCT00850928
Title: Postoperative Cognitive Decline, Inflammation, and Plasma Levels of Beta-amyloids.
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: H08-658
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Postoperative Cognitive Dysfunction; Mild Cognitive Impairment
Keywords: Postoperative Cognitive Dysfunction; MCI; Mild Cognitive Impairment; Aβ40; Aβ42; Apolipoprotein E; Inflammatory Markers; Apolipoprotein E Profile; Serum Beta Amyloid Profile; Inflammatory Markers Profile
MeSH Terms: conditions — Postoperative Cognitive Complications; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma will be collected and stored at baseline, intra-operatively, and one day post-operative for analysis of markers of inflammation. Plasma will be collected and stored at baseline, three months, and six months for analysis of Beta Amyloid levels. DNA will be collected and stored at baseline for analysis of Apolipoprotein E.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects: 65 years and older scheduled for spine surgery will be undergoing serial assessments preoperatively and postoperatively over 6 time-points.

SUMMARY:
Postoperative cognitive dysfunction (POCD) can be a serious complication. The development of therapeutic strategies for the prevention and treatment of this condition requires the identification of subgroup of patients with the greatest incidence of POCD. Several retrospective analyses have raised the possibility that surgery is a risk factor for the accelerated progression of Alzheimer's disease (AD). Moreover, there is increasing evidence that inflammatory mechanisms are involved in the pathogenesis of AD. Major surgery can be associated with a profound systemic inflammatory response. Consequently, it is reasonable to suggest that there is a link between major surgery and the postoperative development of AD in patients who are already at high risk for this complication, e.g. the elderly with mild cognitive impairment. In addition, there are several laboratory investigations that suggest that anesthetic agents increase amyloid peptide levels as well as enhance oligomerization of these proteins. The significance of these findings, however, is unknown. This clinical study seeks to correlate perioperative inflammatory responses, perioperative changes in amyloid-beta protein levels (markers of AD) with neurocognitive and functional outcome in the elderly who are at risk for POCD. This knowledge does not exist, but is essential in the effort to plan perioperative care that can reduce the incidence of POCD as well as improve functional recovery.

DETAILED DESCRIPTION:
We will recruit 50 patients 65 years and older scheduled for spine surgery. The design utilizes prospective serial assessments. The enrolled 50 surgical subjects will be evaluated preoperatively and postoperatively over 6 time-points (preoperatively, inta-op, post op day 1, post op day 7, three months and six months) using a widely accepted set of neurocognitive tests, multiple indices of functional recovery, as well as blood tests for plasma biomarkers of inflammation and β-amyloids. Enrollees will be divided in 2 groups: 25 patients with mild cognitive impairment (diagnosed by clinical assessment) and 25 normal elderly patients.

The definition of normal elderly includes: 1). Global Deterioration Scale (GDS) < 3 and Mini-Mental Exam Score (MMSE) >27; 2). Performance on neurocognitive testing (including memory) that is within 1.5 Standard Deviation (SD) of the age matched normative data; 3). The informant interview confirming no functional impairment in the subject. The definition of MCI includes: self-reported memory and functional complains, a history of memory decline with functional changes that are corroborated by a knowledgeable informant, and a clinical interview resulting in a GDS=3 or higher and MMSE=26 or lower.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 65 and older scheduled to undergo spine surgery.
2. Subjects who are able to read and understand English

Exclusion Criteria:

1. Emergent nature of the procedure which might preclude the conduct of preoperative cognitive examination
2. Participation in any other investigational intervention or clinical study
3. History of psychiatric illnesses (except depression)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 65 years and older scheduled for major spinal surgery.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To examine the effect of surgery on the progression of AD in a population at high risk for this disease through measures of Amyloid Beta levels (AB40 and AB42). levels | 2 years

SECONDARY OUTCOMES:
To determine whether major surgery induces an increase in plasma Aβ40 and Aβ42. | 2 years
To determine whether the pattern of plasma inflammatory markers is different in patients with MCI compared to patients without MCI. | 2 years
To determine whether the Apolipoprotein E genotype correlates with POCD. | 2 years
To examine the relationship between plasma levels of Aβ40 / Aβ42 and subject performance on neurocognitive testing. | 2 years
To establish a correlation between preoperative mild cognitive impaired (MCI) and post operative cognitive decline ( POCD) using neurocognitive testing. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Germaine Cuff, PhD, Study Director — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No